CLINICAL TRIAL: NCT05914987
Title: Profile-Related Evidence Determining Individualized Cancer Therapy in Pancreatic Cancer (PREDICT-PANC)
Brief Title: Determining Individualized Cancer Therapy in Pancreatic Cancer
Acronym: PREDICT-PANC
Status: Recruiting | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Mandana Kamgar, MD, Assistant Professor, Medical College of Wisconsin
Other Study IDs: PRO00048019
Record Dates: First submitted 2023-06-14; First posted 2023-06-22 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Pancreatic Neoplasms
Keywords: Mutation; Genomics; Targeted Therapy; Cancer; Pancreas
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Targeted Therapy — Approved interventions based on the subject's genomic profile will be provided to investigators for consideration for anti-tumor therapy.

SUMMARY:
This is a non-therapeutic exploratory observational precision oncology study designed to collect and analyze data that demonstrate the clinical efficacy and tolerability of personalized treatments based on molecular tumor profiling assessments (i.e., matched therapy) in adult pancreatic cancer patients. Patient medical records, obtained both retrospectively and prospectively, will be examined for results of molecular profiling obtained through standard of care testing to help understand how well molecular testing might predicts response to therapy. Patient demographic and outcome parameters to be evaluated include, but are not limited to, tumor response, time to treatment failure, patient survival, and toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Pathologically confirmed pancreatic cancer.
* Ability to understand a written informed consent document and the willingness to sign it

Exclusion Criteria:

* Age <18 years.
* Primary cancer diagnosis other than pancreatic cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be selected from individuals seeking treatment for pancreatic cancer who have had next generation genomic sequencing of their tumors.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-12-04 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2033-08-01 (Estimated)

PRIMARY OUTCOMES:
Number of Subjects Receiving Targeted Therapy | 5 years
  This measure is the number of study subject's whose treating physician prescribes and subsequently receives the therapeutic recommendation of the Molecular Tumor Board.

CONTACTS AND LOCATIONS:
Overall Officials: Mandana Kamgar, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No